CLINICAL TRIAL: NCT01696916
Title: Development of the Partial Pressure of Carbon Dioxide During 6-min Walking Test and at Night in Patients With Chronic Obstructive Pulmonary Disease IV
Brief Title: Development of the Partial Pressure of Carbon Dioxide During Exercise and at Night in Patients With Chronic Obstructive Pulmonary Disease (COPD) IV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schön Klinik Berchtesgadener Land (Other)
Responsible Party: Principal Investigator, Klaus Kenn, Head physician (department of pneumology), Schön Klinik Berchtesgadener Land
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Sentec2012
Record Dates: First submitted 2012-02-21; First posted 2012-10-02 (Estimated); Last update posted 2014-04-15 (Estimated); Status verified 2014-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; carbon dioxide; 6-minute walking test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- exercise testing (Experimental): 6-minute walking test with pCO2 and pO2 measurement
  Interventions: Procedure: 6-minute walking test

INTERVENTIONS:
Procedure: 6-minute walking test — submaximum exercise test

SUMMARY:
The aim of this study is to investigate the development of partial pressure of carbon dioxide during the 6-min walking test and during night in Chronic Obstructive Pulmonary Disease (COPD)-patients (GOLD stage IV). Therefore the partial pressure of carbon dioxide, oxygen saturation and the heart rate are registered by a device called "Sentec" during the mentioned periods. In addition a measurement of activity is realised by an activity monitor ("Sensewear").

ELIGIBILITY:
Inclusion Criteria:

* COPD IV with and without a respiratory insufficiency
* maximal paCO² of 55mmHg at admission (taken at rest by blood gas analysis without LTOT)

Exclusion Criteria:

* paCO² > 55mmHg
* non-invasive ventilation
* acute exacerbation

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Increase of PaCO2 more than 5mmHg | From time of starting 6-minute walking test until the time of PaCO2-increase of more than 5mmHg assessed up to 6 minutes.

SECONDARY OUTCOMES:
Change of PaCO2 | From the beginning of the 6-minute walking test until peak PaCO2, assessed up to 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Kenn, Dr. med., Study Chair — Klinikum Berchtesgadener Land, Schön Klinik
Locations (1):
- Klinikum Berchtesgadener Land, Berchtesgaden, Germany